CLINICAL TRIAL: NCT04623021
Title: An Open-label, Randomized, Multicenter, Controlled Clinical Trial to Evaluate the Efficacy and Safety of CKD-314 (Nafabelltan) in Hospitalized Adult Patients Diagnosed With COVID-19 Pneumonia
Brief Title: A Study Evaluating the Efficacy and Safety of CKD-314 (Nafabelltan) in Hospitalized Adult Patients Diagnosed With COVID-19 Pneumonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A108_02CVD2014
Record Dates: First submitted 2020-11-05; First posted 2020-11-10 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — nafamostat

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Standard of Care Treatment for COVID-19 Infection
- Nafamostat + Standard of Care (Experimental): Nafamostat mesylate on top of standard of care
  Interventions: Drug: Nafamostat Mesilate

INTERVENTIONS:
Drug: Nafamostat Mesilate — Administered intravenously as a continuous infusion
  Arms: Nafamostat + Standard of Care

SUMMARY:
The primary objective of this study is to evaluate the efficacy of CKD-314 (Nafabelltan) compared to standard of care (SOC), with respect to clinical status assessed by a 7-point ordinal scale in hospitalized adult patients diagnosed with COVID-19 pneumonia

ELIGIBILITY:
Inclusion Criteria:

* Men and women Aged ≥18 years
* Hospitalized subjects who have confirmed COVID-19 infection and have evidence of pneumonia:
* Subjects who are eligible for diagnosis/evaluation to chest X-ray or chest CT
* Women of childbearing potential (including women in post menopause for less than 2 years) must use a medically acceptable forms of birth control and agree to continue its use during the study
* Subjects (or legally authorized representative) should be able to understand and agree to comply with the clinical trial and to provide a written consent document prior to initiation of any study procedure

Exclusion Criteria:

* Subjects who have a record of HIV or AIDS
* Subject has a serious chronic disease
* Active bleeding or ongoing clinical condition deemed at high risk of bleeding contraindicating anticoagulant treatment
* Pregnant or lactating females
* Subjects with liver cirrhosis whose Child-Pugh score is B or C
* Subjects who have liver disease abnormalities with ALT or AST > 5 times ULN
* Estimated glomerular filtration rate (eGFR) < 30 ml/min (including patients receiving hemodialysis or hemofiltration)
* QTcB or QTcF >500ms
* Subjects who have clinically significant ventricular arrhythmias (ventricular tachycardia, ventricular fibrillation) in medical history
* Subjects with rapidly deteriorating clinical condition or low likelihood to complete the study according to the investigator's opinion
* Subjects who are not appropriate for the study, as the investigator's opinion
* Subjects who have hypersensitivity to the investigational drug
* Subjects participated in any other clinical trial (including drugs for the treatment of COVID-19) 3 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
Time to clinical improvement | up to 28 days
  Time to clinical improvement (TTCI) was defined as time (days) from randomization to a decline of 2 categories on the seven-category ordinal scale of clinical status or live discharge from the hospital, whichever came first

SECONDARY OUTCOMES:
Time to recovery | up to 28 days
  Day of recovery is defined as the first day on which the subject satisfies one of the following: 1) Not hospitalized with resumption of normal activities; 2) Not hospitalized, but unable to resume normal activities; 3) Hospitalization, not requiring supplemental oxygen- no longer required ongoing medical care
Proportion of patients with clinical improvement as defined by live discharge from hospital or a decline of 2 categories on the seven-category ordinal scale of clinical status | Day 4, 7, 11, 14 and 28
Proportion of patients with recovery as defined as the subject satisfies one of the following | Day 4, 7, 11, 14 and 28
  1) Not hospitalized with resumption of normal activities; 2) Not hospitalized, but unable to resume normal activities; 3) Hospitalization, not requiring supplemental oxygen- no longer required ongoing medical care
Change of clinical status assessed by 7-category ordinal scale | Day 4, 7, 11, 14 and 28
Change in National Early Warning Score (NEWS) | Day 4, 7, 11, 14 and 28
Time to National Early Warning Score (NEWS) of ≤ 2 which is maintained for 24 hours | up to 28 days
Changes on CT scan/X-ray | Day 5, 11, 14 and 28
  Measured as proportion of patients with improved, not changed or worsened CT scan/X-ray
Change from baseline of CRP | Day 4, 7, 11, 14 and 28
Time to normalize the CRP | up to 28 days
  Decrease to the level of <10 mg/l
Duration of hospitalization | up to 28 days
Duration of non-invasive ventilation or high flow oxygen use | up to 28 days
Incidence of non-invasive ventilation or high flow oxygen use | up to 28 days
  Proportion of patients of non-invasive ventilation or high flow oxygen use
Duration of supplement oxygen use | up to 28 days
Incidence of supplement oxygen use | up to 28 days
  Proportion of patients of supplement oxygen use
Duration of invasive ventilation or extracorporeal membrane oxygenation (ECMO) use | up to 28 days
Incidence of invasive ventilation or extracorporeal membrane oxygenation (ECMO) use | up to 28 days
  Proportion of patients of invasive ventilation or extracorporeal membrane oxygenation (ECMO) use
28-Day mortality | up to 28 days

CONTACTS AND LOCATIONS:
Locations (11):
- Russia (11):
  - A108_02CVD2014 Site# 9, Barnaul
  - A108_02CVD2014 Site# 26, Krasnoyarsk
  - A108_02CVD2014 Site# 5, Moscow
  - A108_02CVD2014 Site# 8, Moscow
  - A108_02CVD2014 Site# 31, Ryazan
  - A108_02CVD2014 Site# 25, Saint Petersburg
  - A108_02CVD2014 Site# 29, Saint Petersburg
  - A108_02CVD2014 Site# 30, Saint Petersburg
  - A108_02CVD2014 Site# 3, Saint Petersburg
  - A108_02CVD2014 Site# 4, Saint Petersburg
  - A108_02CVD2014 site#1, Ufa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhuravel SV, Khmelnitskiy OK, Burlaka OO, Gritsan AI, Goloshchekin BM, Kim S, Hong KY. Nafamostat in hospitalized patients with moderate to severe COVID-19 pneumonia: a randomised Phase II clinical trial. EClinicalMedicine. 2021 Nov;41:101169. doi: 10.1016/j.eclinm.2021.101169. Epub 2021 Oct 27. PMID 34723164